CLINICAL TRIAL: NCT02216721
Title: The Effect of Disease-specific Treatment on Bone Turnover Markers in Patients With Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Principal Investigator, Dr Huai Heng, Loh, Dr, University Malaysia Sarawak
Other Study IDs: FF-2014-267
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Primary Aldosteronism
Keywords: bone mineral density; bone turnover markers; primary aldosteronism treatment
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non primary aldosteronism: Non primary aldosteronism patients undergoing usual anti hypertensive treatment
- Primary Aldosteronism: Patients with confirmed primary aldosteronism undergoing treatment

SUMMARY:
Primary aldosteronism (PA) is a disorder of the adrenal gland causing an autonomous overproduction of mineralocorticoids, leading to arterial hypertension. Although rare, it is the most frequent cause of secondary hypertension. Early detection is important to avoid end organ damage, specifically cardiovascular and metabolic morbidity. Recent studies showed a positive correlation between patients with PA with lower bone density especially at the spine, with significant improvement post treatment, either medically or surgically. There was also a positive correlation between high aldosterone renin ratio with higher levels of intact parathyroid hormone (iPTH) which is responsible for cortical bone loss especially at the distal forearm.

We hypothesize that our patients with PA have a higher level of iPTH, with lower bone density especially at the distal forearm, with improvement post treatment.

DETAILED DESCRIPTION:
In 2004, through an animal model study, rats given aldosterone/salt treatment were found to have reduction in bone mineral density (BMD) and cortical bone strength. This was believed to be due to hypermagnesuria and hypercalciuria leading to bone loss.

This led to subsequent studies which found the association between PA with low serum ionized calcium, increased urine calcium and magnesium, raised intact parathyroid hormone (PTH) levels with subsequent low bone mineral density.

In one small study of 11 patients with confirmed PA taken from a cohort of 188 patients with adrenal incidentaloma, BMD of vertebral, total and neck of femur was found to be lower than non-PA patients, with a higher prevalence of vertebral osteoporotic fractures (72.7% among PA patients vs 20% among non-PA patients). Serum PTH was significantly higher in PA group compared to non-PA group. Six months of treatment either medically or surgically led to significant decrease of urinary calcium excretion and PTH in PA group. Lumbar spine BMD showed significant improvement one year after treatment in 5 patients.

The cross-sectional and interventional data from the GECOH study, which was conducted in a tertiary center in Austria on patients confirmed to have PA, looked at differences in PTH levels between patients with PA (n=10) and essential hypertension (EH) (n=182) and found PTH levels to be significantly higher in PA patients compared with EH group. Treatment with either adrenalectomy or mineralocorticoid receptor antagonists led to a significant decrease of PTH concentrations. Both of these studies had no significant differences in serum Vitamin D level in both cases and controls, as well as pre and post treatment for PA patients. However in the latter study, PTH reduction was found to be more significant in PA patients who underwent adrenalectomy compared to patients treated medically with mineralocorticoid receptor antagonists.

A recent large-scale study on more than 3000 German general adult population showed a significant but non linear association between aldosterone-renin ratio with plasma PTH concentrations, especially in subjects with ARR>90th percentile, despite normal Vitamin D levels. This was believed to be due to the presence of parathyroid receptors type 1 in the adrenals as well as the parathyroid glands expressing mineralocorticoid receptors. However, calcium intake status as well as calcium levels were not assessed in this study.

This findings were all echoed in a few other studies which showed a positive association between PTH levels with PA which was not affected by Vitamin D status.

It is well known that high PTH level is associated with low bone mass and higher osteoporotic fracture risk due to the stimulation effect of PTH on the osteoclastic and osteoblastic activity of the bones resulting in the release of calcium and phosphate from the bone.

Up to date, to our knowledge, there has been no study on the association between PA with bone turnover markers. The use of this sensitive marker as a surrogate indicator of improvement in bone mass pre and post treatment in patients with PA either medically or surgically is novel. The relationship between calcium intake in the patients with the bone metabolism and blood parameters were not looked into previously. In addition, the involvement of peripheral cortical bone mass (distal radius), which is usually associated with elevated PTH, in this group of patients has not been studied.

In this study, we aim to:

1. Assess the BMD of vertebrae, total and femoral neck, and distal third radius in PA patients compared to non-PA.
2. Evaluate the effect of specific treatments on bone turnover markers and BMD in patients with PA
3. Assess the relationship between BMD and bone turnover markers with serum iPTH, calcium, magnesium and vitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Confirmed primary aldosteronism with following criteria i) Aldosterone-renin ratio > 555 SI or 30 (if aldosterone is taken in pmol/L, renin in ng/dL) and ii) Aldosterone post fludrocortisone suppression test > 166pmol/L or >6ng/dL, or iii) Aldosterone post saline suppression test >277pmol/L or >10ng/dL

Exclusion Criteria

1. Patients on medication affecting bone metabolism, eg bisphosphonates, hormonal replacement therapy, SERM, testosterone, antiandrogen, anticonvulsants, calcium and Vitamin D
2. Primary aldosteronism post treatment (surgically or medically on spironolactone or eplerenone)
3. Estimated GFR <30ml/min
4. Severe hepatic failure
5. Severe heart failure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study conducted in out-patient clinics of a tertiary care center. The study population consists of patients referred to our centres for endocrine hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 3 months
  Change of bone mineral density 3 months post treatment for primary aldosteronism

SECONDARY OUTCOMES:
Bone turnover markers | 3 months
  Change of bone turnover markers 3 months post treatment for primary aldosteronism

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Kebangsaan Malaysia, Kuala Lumpur, WP Kuala Lumpur, Malaysia